CLINICAL TRIAL: NCT02895113
Title: Effect of Aspirin on Renal Disease Progression in Patients With Type 2 Diabetes: a Multicentre Double-blind, Placebo-controlled, Randomised Trial. The LEDA (renaL disEase Progression by Aspirin in Diabetic pAtients) Study.
Brief Title: Aspirin and Renal Disease Progression in Patients With Type 2 Diabetes
Acronym: LEDA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Violi, Full professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEDA study
Record Dates: First submitted 2016-09-04; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes
Keywords: Aspirin; Diabetes; Renal function; Thromboxane
MeSH Terms: conditions — Diabetes Mellitus | interventions — Aspirin

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Experimental): Patients will be treated with aspirin 100 mg/day for one year
  Interventions: Drug: Aspirin
- Placebo (Placebo Comparator): Patients will be treated with placebo for one year
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aspirin — Patients suffering from type 2 diabetes will be randomized to receive 100 mg/day or placebo for one year
  Other Names: Cardioaspirin; Acetylsalicylic acid
  Arms: Aspirin
Other: Placebo — Patients in this arm will be treated with placebo
  Arms: Placebo

SUMMARY:
The pathophysiology of diabetes is multifactorial. Beyond genetic susceptibility loci, a lot of acquired risk factors are involved in the development and progression of the disease. Chronic complications of diabetes can be divided into vascular and nonvascular. The risk of developing complications increases with the duration of hyperglycemia, and usually become apparent in the second decade of hyperglycemia. Vascular complications are further subdivided into microvascular (retinopathy, nephropathy and neuropathy) and macrovascular (coronary artery disease, peripheral arterial disease, cerebrovascular disease). It is estimated that the annual decline of estimated glomerular filtration rate (eGFR) in diabetic adults is about 2.1-2.7 ml/min.

While there is consolidated evidence about the use of aspirin (ASA) for secondary prevention in diabetic patients, there is no consensus on the use in primary prevention; the use of ASA in these patients is at physician discretion.

ASA is an effective antithrombotic agent that inhibits the production of thromboxane (Tx) A2 and other prostaglandins by blocking cyclooxygenase (COX). In patients treated with aspirin, serum TxB₂ level is the most reliable in vivo indicator of COX-1 inhibition than TxA2, due to its short half-life and artifacts associated with platelet activation ex vivo.

COX are present in the kidney in the macula densa, in the medulla and in the interstitium. Experimental animals models have demonstrated that COX are involved in regulation of renal blood flow. In particular, in a murine animal model, after the administration of COX inhibitors such as aspirin and celecoxib, it was observed an improvement in renal plasma flow and eGFR, suggesting a role for Tx in the progression of renal damage However, data on the relationship between aspirin and renal function in humans are scarce. In a recent work lead on a large cohort of 800 patients with non-valvular atrial fibrillation, ASA use was associated with a reduced progression of eGFR <45 ml/min during 2 years of follow-up. Furthermore, basal levels of urinary excretion of TxB2, correlated inversely with the use of aspirin and with the decrease of eGFR at follow-up.

The aim of the study is to evaluate the decline in renal function in diabetic patients treated with low-dose aspirin (100 mg/day) vs. untreated diabetic patients.

DETAILED DESCRIPTION:
Epidemiological data show that type 2 diabetes has an epidemic trend worldwide. The increase in food intake, the greater availability of refined grains and the reduction of physical activity had, in fact, negative effects in most areas. It is expected that the number of people suffering from diabetes will double in the period 2000-2030.The most important increase is expected in developing countries, where the prevalence of obesity has rapidly increased. Unlike developing countries, in Europe and in US the higher incidence of diabetes is primarily related to the increased life expectancy of the general population and of diabetic people in particular, and secondary to the higher incidence of the disease. The Casale Monferrato Study indicate an increase of 44% (2.6% vs. 3.8%) in the period 1988-2000. The prevalence of obesity in diabetic patients (Body Mass Index, BMI> 30 kg / m2) increased from 23% to 34%. Whereas in subjects aged <65 years the increase in the prevalence of type 2 diabetes was non-significant (1.1% vs. 1.7%), in the age group > 65 years, the increase was significant (6.5% vs. 9.1%). In particular, a doubling of the prevalence in the age ≥80 years was recorded (3.5% vs. 7.2%). The most recent data from the Turin Study show that in 2003 the prevalence of overt diabetes was 4.9% in 2003. Thus, there was a doubling of cases over a period of 15 years (1988-2003); in the age group 65-74 years, the prevalence rose to 13% and in the age> 74 years to 14%. It is also estimated that 1.5-2% of the population is affected by misdiagnosed diabetes.

The pathophysiology of diabetes is multifactorial. Beyond genetic susceptibility loci, a lot of acquired risk factors are involved in the development and progression of the disease. The most important are Impaired Fasting Glucose (IFG) (odds ratio, OR = 11), Impaired Glucose Tolerance (IGT) (OR = 3.9), the weight (overweight: OR = 3.4 and obesity: OR = 9.9), dyslipidemia (OR = 1.6), hypertension (OR = 2.3).

Chronic complications of diabetes can be divided into vascular and nonvascular. The risk of developing complications increases with the duration of hyperglycemia, and usually become apparent in the second decade of hyperglycemia. Vascular complications are further subdivided into microvascular (retinopathy, nephropathy and neuropathy) and macrovascular (coronary artery disease, peripheral arterial disease, cerebrovascular disease). In particular, the worsening of renal function seems to be a peculiar characteristic of the patients suffering from diabetes. It is estimated that the annual decline of estimated glomerular filtration rate (eGFR) in diabetic adults is about 2.1-2.7 ml/min.

Aspirin and Diabetes The efficacy and the safety of acetylsalicylic acid (aspirin, ASA) as an antithrombotic agent has been assessed in different subsets, both in apparently healthy people at low risk of vascular complications (primary prevention), and in high-risk patients, such as those with a previous myocardial infarction or acute ischemic stroke (secondary prevention). Diabetic patients represent an important group in whom treatment with ASA should be carefully considered. The evidence that type 2 diabetic patients taking glucose-lowering agents have similar cardiovascular risk compared to non-diabetic with a previous myocardial infarction, could make reasonable the use of an antiplatelet drug as primary prevention strategy for cardiovascular diseases. However, while there is consolidated evidence about the use of ASA for secondary prevention in diabetic patients, there is no consensus on the use in primary prevention; ASA use in these patients is at physician discretion.

Mechanism of action of aspirin. Aspirin is an effective antithrombotic agent that inhibits, the production of thromboxane (Tx) A2 and other prostaglandins by blocking cyclooxygenase (COX) enzyme. There have been described two isoforms of COX, the COX-1, which is widely expressed and which plays a function of gastric cyto-protection, and COX-2 expressed upon external stimuli and mainly in inflammatory and immune cells. Low-dosage ASA can inhibit COX-1, while at high dosage, ASA can inhibit both COX-1 and COX-2 enzymes.

The antiplatelet action of ASA is via specific inhibition of COX in platelets, through the acetylation of serine-529 of COX-1. This enzyme possesses both cyclooxygenase activity [converting arachidonate into prostaglandin G2 (PGG2)] and peroxidase [converting PGG2 into PGH2, the biochemical precursor of many other prostaglandins and Tx]. In platelets, this inhibitory effect has as a result, the reduced production of prostaglandins and TxA2, which is a strong platelet agonist. This inhibitory effect is irreversible so that TxA2-mediated platelet aggregation can be restored only through the synthesis of new platelets. Thus, after ASA administration, platelet aggregation is inhibited up to 7 days.

In patients treated with low doses of aspirin, serum TxB₂ level is a most reliable in vivo indicator of COX-1 inhibition than TxA2, due to its short half-life and artifacts associated with platelet activation ex vivo.

Both urinary levels of 11-dehydro-TxB₂ and 2.3-dinor-TxB₂, the most abundant metabolite of TxB₂, have been proven to be platelet activation surrogates. As 11-dehydro-TxB₂ is excreted in higher amounts and has a longer half-life, is the marker of choice.

Thromboxane binds to TP receptor, commonly found on platelets, smooth muscle cells, endothelium and vessels. They exert vasoconstriction function on blood vessels, platelet aggregation and induce the initial stages of coagulation. In particular, Tx is entailed in the reduction of renal blood flow and glomerular filtration rate.

Optimal dosage of aspirin. Randomized placebo-controlled studies have shown that aspirin is effective as an antithrombotic agent at a dosage ranging from 50 to 1500 mg/day; however, long-term clinical efficacy requires daily dosage of 50 up to 100 mg/day.

Patrono et al. assessed a relationship between aspirin dose and TxB2 levels. This study showed that a single dose of 100 mg of drug was able to reduce by 98% the concentration of serum levels of Tx during the first hour. Single doses of 100-400 mg were able to reduce of 94-98% after 24 and 48 hours, with an inhibition rate up to 90-92% at 72 hrs. Serum Tx decreased to normal levels after a period compatible with the platelet half-life. More than 90% of platelet inhibition could be maintained over one month by giving 200 mg of aspirin every 72 hours.

Aspirin, eicosanoids and renal function As previously reported, ASA is able to inhibit Tx production by inhibiting COX; COX are present in the kidney in the macula densa, in the medulla and in the interstitium. In the macula densa this enzyme seems to favour renin production (eg. salt restriction, use of ACE inhibitors, renovascular hypertension).

Experimental animals models have demonstrated that COX are involved in regulation of renal blood flow. In particular, in a murine animal model, after the administration of COX inhibitors such as aspirin and celecoxib, it was observed an improvement in renal plasma flow and eGFR, suggesting a role for Tx in the progression of renal damage.

However, data on the relationship between aspirin and renal function in humans are not available. In a recent work that included a large cohort of 800 patients with non-valvular atrial fibrillation, the use of aspirin was associated with a reduced progression of eGFR <45 ml/min during 2 years of follow-up. In particular, patients not receiving aspirin had an incidence of GFR <45 ml/min of 15% vs. 5% of those treated with aspirin 100 mg/day. Furthermore, basal levels of urinary excretion of TxB2, correlated inversely with the use of aspirin and with the decrease of eGFR at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes: random blood glucose ≥ 200 mg / dl, fasting blood glucose ≥ 126 mg/dl, blood glucose 2 hours after oral glucose tolerance test (75 g) ≥200 mg/dl, treatment with glucose-lowering agents.

Exclusion Criteria:

1. History of cardiovascular or cerebrovascular events;
2. Presence of inadequate glycaemic control (glycosylated haemoglobin ≥8%);
3. Clinical diagnosis of type 1 diabetes (diagnosis of diabetes and insulin use before 35 years of age);
4. Patients with renal impairment in G4 stage (eGFR <30 ml/min) at baseline;
5. Chronic active infection or evidence of malignancy in the last 5 years;
6. Autoimmune systemic disease;
7. Cardiac arrhythmia;
8. Use of non-steroidal anti-inflammatory drugs, vitamin supplements, or other antiplatelet agents in the previous 30 days;
9. Liver Failure (eg cirrhosis);
10. Use of anticoagulants;
11. Life expectancy <1 year;
12. Known allergy to aspirin.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Changes in renal function in diabetic patients treated with aspirin | 1 year
  The aim of our study is to evaluate the decline in renal function in diabetic patients treated with low-dose aspirin (100 mg/day) vs. untreated diabetic patients. In particular, we will evaluate:
  * The absolute change in eGFR, calculated as the difference between eGFR at 12 months - baseline eGFR;
  * The rapid decline in renal function, defined as a reduction of eGFR ≥5 ml/min at 1 years.
  * The change of renal function class (from G1 to G2, from G2 to G3a and so on) at 6 and 12 months.

SECONDARY OUTCOMES:
Relationship between changes of Thromboxane B2 excretion and renal function in diabetic patients treated with aspirin | 1 year
  As secondary endpoint, we will evaluate changes in the urinary excretion TxB2 both baseline and at one year. Changing levels of urinary TxB2 will then be related to renal function.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Violi, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Internal and Medical Specialities Department - Policlinico Umberto I, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715
- [Background] Davi G, Patrono C. Platelet activation and atherothrombosis. N Engl J Med. 2007 Dec 13;357(24):2482-94. doi: 10.1056/NEJMra071014. No abstract available. PMID 18077812
- [Background] Patrono C, Ciabattoni G, Pinca E, Pugliese F, Castrucci G, De Salvo A, Satta MA, Peskar BA. Low dose aspirin and inhibition of thromboxane B2 production in healthy subjects. Thromb Res. 1980 Feb 1-15;17(3-4):317-27. doi: 10.1016/0049-3848(80)90066-3. No abstract available. PMID 7368167
- [Background] Lariviere R, Moreau C, Rodrigue ME, Lebel M. Thromboxane blockade reduces blood pressure and progression of renal failure independent of endothelin-1 in uremic rats. Prostaglandins Leukot Essent Fatty Acids. 2004 Aug;71(2):103-9. doi: 10.1016/j.plefa.2003.12.021. PMID 15207526
- [Background] Lomnicka M, Karouni K, Sue M, Wessel LA, Bing RJ. Effects of nonsteroidal anti-inflammatory drugs on prostacyclin and thromboxane in the kidney. Pharmacology. 2003 Jul;68(3):147-53. doi: 10.1159/000070172. PMID 12784086
- [Background] Pastori D, Pignatelli P, Perticone F, Sciacqua A, Carnevale R, Farcomeni A, Basili S, Corazza GR, Davi G, Lip GYH, Violi F; ARAPACIS (Atrial Fibrillation Registry for Ankle-Brachial Index Prevalence Assessment-Collaborative Italian Study) study group. Aspirin and renal insufficiency progression in patients with atrial fibrillation and chronic kidney disease. Int J Cardiol. 2016 Nov 15;223:619-624. doi: 10.1016/j.ijcard.2016.08.224. Epub 2016 Aug 14. PMID 27565838
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Violi F, Targher G, Vestri A, Carnevale R, Averna M, Farcomeni A, Lenzi A, Angelico F, Cipollone F, Pastori D. Effect of aspirin on renal disease progression in patients with type 2 diabetes: A multicenter, double-blind, placebo-controlled, randomized trial. The renaL disEase progression by aspirin in diabetic pAtients (LEDA) trial. Rationale and study design. Am Heart J. 2017 Jul;189:120-127. doi: 10.1016/j.ahj.2017.04.005. Epub 2017 Apr 18. PMID 28625368